CLINICAL TRIAL: NCT07143097
Title: Effect of Capecitabine as Maintenance Therapy Versus Observation on Patients With Early Stage Triple Negative Breast Cancer
Brief Title: Capecitabine as Maintenance Therapy vs Observation in Early-stage Triple-negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sarah Hamdy Ali Sayed, assistant lecturer of clinical oncology, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC/10102021/Sayed
Record Dates: First submitted 2025-08-09; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Triple -Negative Breast Cancer
Keywords: early stage breast cancer triple negative
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- receive low-dose capecitabine maintenance within 4 weeks of finishing the standard adjuvant tr (Experimental)
  Interventions: Drug: capecitabine
- No Intervention: observation after finishing the standard adjuvant treatment (No Intervention)

INTERVENTIONS:
Drug: capecitabine — capecitabine 650 mg / m2 twice per day for one year
  Other Names: xeloda
  Arms: receive low-dose capecitabine maintenance within 4 weeks of finishing the standard adjuvant tr

SUMMARY:
Eligible patients was assigned in a 1:1 ratio to receive either low-dose capecitabine maintenance (intervention group) which is newly diagnostic to be planned to receive capecitabine after finishing the standard adjuvant treatment or observation (control group) within 4 weeks after completion of standard adjuvant chemotherapy.

DETAILED DESCRIPTION:
Eligible patients will randomly open label assigned in a 1:1 ratio to receive either low-dose capecitabine maintenance (intervention group) which is newly diagnostic to be planned to receive capecitabine after finishing the standard adjuvant treatment or observation (control group) within 4 weeks after completion of standard adjuvant chemotherapy.

The capecitabine maintenance group will receive oral capecitabine at 650 mg/m2, twice daily continuously for 1 year.

Total follow up of the study is 2 years, one year for drug receving with monthy follow up for adverse effect and the other year for every 3 months follow up to asses DFS and OS.

Collection of capecitabine dose will receive and adverse events will assessed monthly during capecitabine maintenance in the capecitabine group. In both groups, physical examination, assessment of menopausal status, breast ultrasound, and abdominal ultrasound were performed every 3 months during 2 years of follow up; mammography and chest x-ray were performed yearly. Patients who has not experienced recurrence or death at the time of data analysis will censored as alive and event-free at the date of last follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Eligible trial participants will women who has pathologically confirmed invasive breast ductal carcinoma Hormone receptor negative (<1% positive cells by immunohistochemistry staining) and ERBB2 negative.

Participants had early-stage tumors that were stage T1b-3N0-3cM0, without positive supraclavicular or internal mammary lymph node.

They received standard treatments, including modified radical mastectomy or breast-conserving surgery, neo-/adjuvant chemotherapy, and radiotherapy according to institutional guidelines.

* patients were able to swallow tablets
* performance status 0 - 1

Exclusion Criteria:

* Key exclusion criteria will include Inflammatory or bilateral breast cancer. History of invasive breast cancer or other malignancies; receipt of other biologic agents or immunotherapy.

Lactation or pregnancy; or severe coexisting illness.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
adverse effents of capictabine | assess the adverse effects of the Capecitabine 6 months after starting treatment.

SECONDARY OUTCOMES:
distant disease-free survival | up to 24 months from diagnosis
  defined as the time from randomization to the first occurrence of the following events: local relapse, distant metastasis or contralateral breast cancer.
overall survival | 24 months from diagnosis
  the time from randomization to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Eligible patients will randomly in a 1:1 ratio to receive either low-dose capecitabine maintenance (intervention group) which is newly diagnostic to be planned to receive capecitabine after finishing the standard adjuvant treatment or observation (control group) within 4 weeks after completion of standard adjuvant chemotherapy.
  The capecitabine maintenance group will receive oral capecitabine at 650 mg/m2, twice daily continuously for 1 year.
Supporting Information: Study Protocol, SAP
Time Frame: Total follow up of the study is 2 years, one year for drug receving with monthy follow up for adverse effect and the other year for every 3 months follow up to asses DFS and OS.
Access Criteria: for oncologists

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT07143097/Prot_SAP_000.pdf